CLINICAL TRIAL: NCT02496286
Title: Feasibility Study of Intraperitoneal Bevacizumab for Palliation of Intractable Malignant Ascites
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Eastern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: EP2014013
Record Dates: First submitted 2015-07-01; First posted 2015-07-14 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Malignant Ascites
Keywords: Necessary paracentesis for symptom control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eligible patients requiring paracentesis for symptom control (Experimental)
  Interventions: Drug: Intraperitoneal Bevacizumab

INTERVENTIONS:
Drug: Intraperitoneal Bevacizumab — Bevacizumab 200mg diluted in 250 ml of normal saline

SUMMARY:
This study will evaluate the safety and efficacy of intraperitoneal administration of Bevacizumab to prevent the recurrence of malignant ascites. Ten patients will receive intraperitoneal Bevacizumab 200 mg in 250 ml of normal saline for infusion every two weeks for up to six weeks, or a maximum of three treatments.

DETAILED DESCRIPTION:
This protocol describes a pilot study to assess whether intraperitoneal Bevacizumab infusion is safe and improves the time to repeat paracentesis. In patients with non-draining malignant peritoneal effusion, published data suggests that the average time to repeat paracentesis in malignant ascites is 10-13 Days. The investigators' treatment will be considered potentially efficacious if the median time to repeat paracentesis is greater than 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the case of:

  * Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2
  * Participants must be 18 years of age or older
  * Have ascites of malignant disease
  * Have symptoms related to ascites
  * Ascites Index above 0.05 (AI ˃ 0.05)
  * Be an English speaking patient or have an interpreter available
  * Be able to understand and comply with all study requirements and the implications of off-label use of intraperitoneal Bevacizumab
  * Have had at least two paracentesis within the last 4 weeks

Exclusion Criteria:

* Patients will be excluded in the case of:

  * Ascites due to non-malignant cause
  * Concurrent treatment with systemic chemotherapy that has a realistic chance of controlling the ascites
  * Concurrent treatment with intraperitoneal Bevacizumab
  * life expectancy of less than 2 weeks
  * A history of bowel perforation or fistula
  * Symptoms or signs suggestive of bacterial peritonitis
  * Child's C cirrhosis
  * Uncontrolled hypertension
  * Surgery within 28 days of catheter treatment
  * Evidence of coagulopathy
  * Symptoms suggestive of bowel obstruction
  * Major surgery, open biopsy or significant traumatic injury within seven (7) days of first study drug--including neurosurgery.
  * Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements.
  * Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements
  * Patients who are pregnant or lactating (females of childbearing potential must have a negative pregnancy test prior to participation)
  * Patients with pre-existing 3 + or greater urine dipstick reading proteinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Radiographic Improvement | 14 days (+/-4 days)
  Radiographic improvement in area of intraperitoneal collection will be evaluated (between the area of the intraperitoneal collection on the ultrasound pre-procedure and ultrasound evaluation on day 14 (+/-4 days).
Volume Output | 14 days (+/-4 days)
  Change in volume output from baseline to day 14 (+/-4 days)

SECONDARY OUTCOMES:
Adverse Events | 14 days (+/-4 days)
  Adverse events will be judged possibly or probably related to intraperitoneal Bevacizumab infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Regional Medical Center, Philadelphia, Pennsylvania, United States